CLINICAL TRIAL: NCT01945918
Title: Comparing Strategies for Translating Self-management Support Into Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of California, San Francisco (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-0645; 1R18DK096387-01 (NIH)
Record Dates: First submitted 2013-08-27; First posted 2013-09-19 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Diabetes Mellitus; Primary Health Care; Self care
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Self-management support education (Active Comparator): Project staff will meet onsite with practice clinicians for a two-hour session to discuss what self-management support (SMS) is, why it is important, how primary care plays a role in this process, how others have approached it, and how it can be time and cost efficient for them to engage in SMS as part of standard diabetes care. Practices will have access to a website displaying general and local SMS resources. Discussion of the implementation of these resources into the practice will be facilitated. Two additional academic detailing visits will be made to check on progress on SMS adoption, provide additional information as needed, and answer questions. No input will be provided regarding how unique practice characteristics might be utilized for more effective implementation of SMS, and CTH will not be introduced.
  Interventions: Behavioral: Self-management support education
- Connection to Health Interactive Behavior Change Technology (Active Comparator): Connection to Health (CTH) Arm: The number and length of staff visits to these practices will be the same as for the SMS Education Arm, but the content of the visits will center on the implementation and use of the CTH program as a way to implement SMS. Clinicians and selected staff members will be given hands-on experience using the system and will be provided with scenarios that will highlight the effective use of CTH as a tool for diabetes SMS. The practices will then implement CTH, using protocols selected from several suggested by the research team. Additional technical assistance with implementing CTH will also be provided as needed.
  Interventions: Behavioral: Connection to Health Interactive Behavior Change Technology
- Connection to Health plus Coaching (Experimental): Connection to Health plus Coaching (CTH+C) Arm: This arm adds practice coaching as described above to CTH. The active coaching phase focuses on meetings of the practice improvement team, scheduled every other week for approximately 40 minutes each. The improvement team will consist of 6 - 10 diverse representatives of the practice (e.g., front office, medical assistants, physicians). The coach will assist the team in developing a CTH adoption plan and then help them break it down into small bites for rapid cycle change using the Plan-Do-Study-Act quality improvement (QI) model. Active coaching will last for 3 months, followed by monthly calls by the coach to review data regarding the practice's use of CTH and brief "booster" coaching to deal with problems.
  Interventions: Behavioral: Connection to Health Interactive Behavior Change Technology; Behavioral: Connection to Health plus Coaching (CTH+C)

INTERVENTIONS:
Behavioral: Self-management support education — Same as Arm Description
  Arms: Self-management support education
Behavioral: Connection to Health Interactive Behavior Change Technology — Same as Arm Description
  Arms: Connection to Health Interactive Behavior Change Technology; Connection to Health plus Coaching
Behavioral: Connection to Health plus Coaching (CTH+C) — Same as Arm Description
  Arms: Connection to Health plus Coaching

SUMMARY:
This project will test different ways of helping primary care practices to do a better job of self-management support (SMS) for their patients with diabetes.

DETAILED DESCRIPTION:
The specific aims of the proposed study are:

* Primary Specific Aims

  1. To conduct a cluster randomized trial to examine the reach, effectiveness, adoption, implementation and maintenance (RE-AIM) of Connection to Health (CTH) for patients with type 2 diabetes in primary care practice settings. Primary effectiveness outcomes will include hemoglobin A1c, Body Mass Index (BMI), blood pressure and Low Desity Lipprotein (LDL) cholesterol.
  2. To determine the incremental benefit, using the RE-AIM framework, of brief targeted practice coaching on the implementation of CTH in diverse primary care practices.
* Secondary Specific Aims

  1. To identify key practice characteristics (e.g., practice size, organization, setting, and level of experience with practice redesign efforts) that impact CTH RE-AIM. These results will inform dissemination of the CTH intervention.
  2. To determine the relative costs associated with implementing CTH and practice coaching to further inform dissemination efforts.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years old or over
* Type 2 Diabetes Mellitus diagnosed for a minimum of 12 months
* Able to read in English or Spanish
* Plan to remain in the practice during the study period

Exclusion Criteria:

* Developmentally disabled
* Decisionally challenged
* Pregnant women

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to 18 months | 18 months from baseline
  Glycosylated hemoglobin (HbA1c) will be measured at baseline and 18 months from baseline.
Change in LDL from baseline to 18 months | 18 months from baseline
  Low-density lipoprotein (LDL) cholesterol will be measured at baseline and 18 months from baseline (in mg/dL; e.g., 160 mg/dL).
Change in systolic and diastolic blood pressure from baseline to 18 months | 18 months from baseline
  Systolic and diastolic blood pressure will be measured at baseline and 18 months from baseline (in mmHg; e.g., 140/90 mmHg)
Change in body mass index (BMI) from baseline to 18 months | 18 months from baseline
  Body mass index (BMI) will be measured at baseline and 18 months from baseline (weight (kg) / [height (m)]2; e.g., 24.96)

SECONDARY OUTCOMES:
Evidence of documented self-management support for patients through medical record review | 18 months from baseline
  The following elements will be assessed in medical record review: presence of a personal care plan with regular updating, evidence of collaborative goal setting, evidence of action planning around prioritized patient goals, evidence of collaborative problem-solving regarding the action planning process, use of community resources to assist in goal attainment, and evidence of ongoing monitoring of progress on identified goals. A total score will be the sum of positive elements.

OTHER OUTCOMES:
Change in patient-reported dietary intake of saturated fat, fruits and vegetables, salt, and sweetened beverages baseline to 18 months | 18 months from baseline
  Patients' dietary intake of saturated fat, fruits and vegetables, salt, and sweetened beverages will be assessed at baseline and 18 months from baseline through a patient-completed survey on their diet.
Change in patient-reported physical activity from baseline to 18 months | 18 months from baseline
  Patients' frequency and duration of participation in vigorous, moderate, and walking activity as well as "screen" time and time spent sitting will be assessed at baseline and 18 months from baseline through a patient-completed survey on their physical activity.
Change in patient-reported tobacco use from baseline to 18 months | 18 months from baseline
  Patients' use of tobacco (whether or not using tobacco, if so, how much; e.g., current smoker [yes/no]; number of cigarettes [10 in the past week]) will be assessed at baseline and 18 months from baseline through a patient-completed survey.
Change in patient-reported medication adherence from baseline to 18 months | 18 months from baseline
  Patients' prescribed medication adherence (number of days missed, reasons for missing) will be assessed at baseline and 18 months from baseline through a patient-completed survey.
Change in patient-reported disease-related distress rating from baseline to 18 months | 18 months from baseline
  Patients' distress related to their diabetes (6-point scales for each item; mean score calculated for each sub-scale [range between 1 and 6]) will be assessed at baseline and 18 months from baseline through a patient-completed survey.
Change in patient-reported diabetes self-care rating from baseline to 18 months | 18 months from baseline
  Patients' measure of the frequency of performing diabetes self-care tasks over the preceding 7 days will be assessed at baseline and 18 months from baseline through a patient-completed survey.

CONTACTS AND LOCATIONS:
Overall Officials: W. Perry Dickinson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver and Health Sciences Center, Aurora, Colorado, United States

REFERENCES:
- [Derived] Hessler DM, Fisher L, Bowyer V, Dickinson LM, Jortberg BT, Kwan B, Fernald DH, Simpson M, Dickinson WP. Self-management support for chronic disease in primary care: frequency of patient self-management problems and patient reported priorities, and alignment with ultimate behavior goal selection. BMC Fam Pract. 2019 Aug 29;20(1):120. doi: 10.1186/s12875-019-1012-x. PMID 31464589
- [Derived] Dickinson WP, Dickinson LM, Jortberg BT, Hessler DM, Fernald DH, Fisher L. A protocol for a cluster randomized trial comparing strategies for translating self-management support into primary care practices. BMC Fam Pract. 2018 Jul 24;19(1):126. doi: 10.1186/s12875-018-0810-x. PMID 30041598